CLINICAL TRIAL: NCT05224700
Title: Early Development of Academic Skills in the Classroom: Short- and Mid-term Effects of a Tablet-based Game That Stimulates Cognitive, Emotional, and Social Skills for Pre-kindergarten Children
Brief Title: Early Development of Academic Skills in the Classroom
Acronym: JAPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Talca (Other)
Collaborators: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Cristián A. Rojas-Barahona, Principal Investigator, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FR 1210989
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: General Population of Children Aged 3 to 5 Years Old
Keywords: cognitive skills; executive function; pre-calculation; literacy learning; emotional skills; social competences

STUDY DESIGN:
Intervention Model Description: Single-blinded, two-arm randomized controlled trial clinical
Who Masked: Outcomes Assessor
Masking Description: In all evaluations, the evaluators will be blind to the trial arm where the schools/students were allocated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The evaluator in charge will monitor the autonomous work of the participants during all 20 sessions of the program for stimulating cognitive and socioemotional skills while also answering questions, training the educators, and solving their doubts about the program and its implementation.
  Interventions: Behavioral: JAPI
- Painting group (Sham Comparator): Each child will play on a tablet with headphones during 20 sessions lasting 30 minutes each, 2 times per week. They will play a tablet-based painting game that involves no cognitive, emotional, or social competence stimulation
  Interventions: Behavioral: Painting group

INTERVENTIONS:
Behavioral: JAPI — Each child will play on a tablet with headphones during 20 sessions lasting 30 minutes each, 2 times per week. All the activities are games with the following structure: an introduction with instructions and protagonist selection, followed by a practice exercise to ensure that the children understand what they have to do (the exercise is repeated until the child performs it correctly), and, finally, the activity itself (4 different activities with 5 tries each). The first 10 sessions jointly stimulate working memory and emotion knowledge (4 activities focused on each skill per session), while the 10 remaining sessions stimulate inhibitory control and the selection of prosocial behaviours. In the inhibitory control activities, they must suppress automatic stimuli and processes; in the emotion recognition activities, they must identify basic emotions; and in the selection of prosocial behaviours, they must choose an option to deal with a social problem.
  Arms: Intervention group
Behavioral: Painting group — Each child will play on a tablet with headphones during 20 sessions lasting 30 minutes each, 2 times per week. They will play a tablet-based painting game that involves no cognitive, emotional, or social competence stimulation
  Arms: Painting group

SUMMARY:
This is a two-arm cluster randomized controlled trial. The two arms will be: 1) Intervention group, where the stimulation program will be implemented; and 2) Comparison group (active).

The aim of this study is: To evaluate the effectiveness of a program aimed at stimulating cognitive (working memory and inhibitory control), emotional (emotion recognition), and social competence skills (choice of prosocial behaviors) for the development of initial literacy learning and pre-calculation in socioeconomically disadvantaged preschoolers immediately after the intervention and at 6, 12, 18, and 24 months post intervention, controlling for gender, mental health, and baseline state of the skills stimulated.

The intervention program, which targets cognitive, emotional, and social competence skills, was designed for socioeconomically disadvantaged preschoolers in order to stimulate their working memory, inhibitory control, emotion recognition, and choice of prosocial behaviors during the development of the academic skills of initial literacy learning and pre-calculation. Immediately after the completion of the intervention program, participants are expected to show improvements in these skills and the academic skills of initial literacy learning and pre-calculation.

DETAILED DESCRIPTION:
General background information:

The literature suggests that children born to low-income families can begin the preschool stage with less developed academic skills (such as pre-calculation and initial literacy learning) and non-academic skills (such as emotional and social competence) compared to children from higher-income families. These differences appear to increase socioemotional, educational, and health-related disparities in the long term. Furthermore, the available evidence indicates that several landmarks of human development take place between 3 and 7 years of age, including the emergence of emotion recognition, control over one's behavior, and executive functions. Therefore, it is essential to work with children who are more economically vulnerable, stimulating these skills at an early age.

Working memory and inhibitory control (executive functions) have been identified as key components in the development of academic skills such as early literacy learning and pre-calculation, with evidence that participants can be stimulated at an early age. Furthermore, a meta-analysis conducted by Blewitt et al. (2018), which examined programs for children aged 2 - 6 years, found that children exposed to social and emotional stimulation programs exhibited significant improvements in social and emotional competences, learning outcomes, and behavioral regulation, while their emotional and behavioral problems were reduced. Several skill-building initiatives aimed at children which involve the use of tactile devices have been reported. For example, Herodotou (2017) conducted a systematic review in order to examine how using tactile screen devices impacted on the learning of children aged 2 to 5 years, finding that most studies evaluated cognitive aspects and largely overlooked socioemotional aspects. However, to the best of our knowledge, no effectiveness evaluations of a program combining cognitive and socioemotional stimulation have been conducted, let alone of a tablet-based program for preschoolers that involves mid-term follow-up.

Specific background information:

Several successful experiences of early cognitive skill stimulation exist, including COGMED for children with ADHD aged 7-17 years (Klingberg et al., 2005) and Memory Booster for children aged 5-8 years (St Clair-Thompson et al., 2010). Examples of socioemotional skill stimulation include PATHS, which involves verbalizing feelings and the usage of self-control strategies. However, our search yielded no effectiveness evaluations of a program combining cognitive and socioemotional stimulation, let alone of a tablet-based program for preschoolers featuring mid-term follow-up. The experience of our research team stems which found results favoring the intervention group in children aged 4-5 years (with a delta greater than 10%), both when stimulating working memory (Rojas-Barahona et al., 2015) and inhibitory control and planning (Rojas-Barahona et al., 2021). The intervention was conducted using a tablet computer in establishments with a high index of school vulnerability (ISV; Spanish: índice de vulnerabilidad escolar, IVE). Therefore, there is evidence in Chile, with socioeconomically disadvantaged preschool-age children, showing that the stimulation of cognitive skills (such as executive functions: working memory and inhibitory control) improves cognitive development and academic skills such as initial literacy learning and pre-calculation. In this context, the aim of this study is to determine the effectiveness of a program that jointly stimulates the cognitive and socioemotional skills of preschoolers in order to boost the development of their academic skills, controlling for gender, mental health, and baseline skills.

Objective of the project:

- To evaluate the effectiveness of a program aimed at stimulating cognitive (working memory and inhibitory control), emotional (emotion recognition), and social competence skills (choice of prosocial behaviors) for the development of initial literacy learning and pre-calculation in socioeconomically disadvantaged preschoolers immediately after the intervention and at 6, 12, 18, and 24 months post intervention, controlling for gender, mental health, and baseline state of the skills stimulated.

Specific objectives Objective 1. To determine the acceptability and ease of use of a program for stimulating cognitive (working memory and inhibitory control), emotional (emotion recognition), and social competence skills (choice of prosocial behaviors) in socioeconomically disadvantaged preschoolers.

Objective 2. To evaluate the changes observed in the variables working memory, inhibitory control, emotion recognition, and choice of prosocial behaviors in both the intervention and the comparison group immediately after the intervention and at 6, 12, 18, and 24 months post intervention.

Objective 3. To determine the effectiveness of a program aimed at stimulating cognitive (working memory and inhibitory control), emotional (emotion recognition), and social competence skills (choice of prosocial behaviors) for the development of initial literacy learning in socioeconomically disadvantaged preschoolers immediately after the intervention and at 6, 12, 18, and 24 months post intervention, controlling for gender, mental health, and baseline state of the skills stimulated.

Objective 4. To determine the effectiveness of a program aimed at stimulating cognitive (working memory and inhibitory control), emotional (emotion recognition), and social competence skills (choice of prosocial behaviors) for the development of pre-calculation in socioeconomically disadvantaged preschoolers immediately after the intervention and at 6, 12, 18, and 24 months post intervention, controlling for gender, mental health, and baseline state of the skills stimulated.

Objective 5. To explore the influence of potential mediators (working memory, inhibitory control, emotion recognition, and choice of prosocial skills) on the observed effects of a program for stimulating cognitive (working memory and inhibitory control), emotional (emotion recognition), and social competence skills (choice of prosocial behaviors), controlling for gender, mental health, and baseline status of the skills stimulated.

Methodology:

Design: A quantitative methodology will be employed, with a two-arm cluster randomized controlled trial design. The two arms will be: 1) Intervention group, where the stimulation program will be implemented; and 2) Comparison group (active). Investigators will establish the explanatory capacity of the independent variables -belonging to the intervention or comparison group- on the dependent variables -development of academic skills (initial literacy learning and pre-calculation)- (main outcome). The team will also consider the following as variables that mediate the effect of the intervention: working memory, inhibitory control, emotion recognition, and ability to select prosocial behaviors. Investigators will perform 1 measurement before the stimulation (pre) and 5 post measurements: immediately after the stimulation and at 6, 12, 18, and 24 months.

Participants: Our sample will comprise co-educational schools that serve preschool-age children located in two cities of the region (Talca and Linares), which have at least two classes per level, and which have an ISV ≥70%. Investigators will randomly select 20 schools in Talca and Linares proportionally to the size of each city's population. Then, schools' principals will be invited to participate. The first 18 institutions that agree will enter the study. The remaining schools that agree to participate will be placed on a waiting list in case any others withdraw from the study or encounter any difficulties (for details, see "Sample size"). Once the schools have been recruited, children will be randomly distributed at a 1:1 ratio through a computerized procedure. A statistician unaffiliated to the research team will conduct the randomization procedure. Afterwards, investigators will invite pre-kindergarten educators and assistants to join the study (together with kindergarten and 1st grade educators, as part of the longitudinal study). Then, during a parent-teacher conference, investigators will invite all the parents and guardians in these classes to allow their children to participate in the study. All three groups of participants (principals, educators and assistants, and parents) will need to sign an informed consent form. All the children authorized to do so will participate in the study; however, the analyses will not consider the data provided by children with cognitive disabilities (with a prior diagnosis). Also, children will need to give their informed assent to participate in the study. Even if their parents have given their consent, any child who does not wish to participate will not be compelled to do so.

Sample size: To determine a significant difference (alpha =0.05) in the measurement of the main result (academic skills: early literacy learning/pre-calculation) between the Comparison and Intervention groups with a statistical power of 80%, the research needs to recruit 6 schools with a total of 264 students per group, with an average of 44 students per school (divided into two classes). Sample size was calculated using the Stata statistical package and the "clustersampsi" command, which makes it possible to identify differences between groups relative to an average score and considers the effect of correlation among subjects within a school by means of the intracluster correlation coefficient. The information used to feed this equation was taken from a prior study (Rojas-Barahona et al., 2015) where the control group, at post-intervention, scored 20.06 for the variable early literacy learning (SD = 8.32). The sample size for this study was calculated assuming a 0.4 SD difference in favour of the intervention group. Estimating that 10% of the eligible students may not want to participate and estimating a 20% loss during follow-up, each group should recruit 377 students initially. This means that the team needs to recruit 9 additional schools per group, for a total of 18 schools.

Description of the groups

-Intervention Group: the intervention will be delivered through a tablet computer game that stimulates cognitive (working memory and inhibitory control), emotional (emotion recognition), and social competence skills (selection of prosocial behaviors). The intervention will be conducted individually in classroom settings; that is, each child will play on a tablet with headphones during 20 sessions lasting 30 minutes each, 2 times per week (2 and a half months in total) (Rojas-Barahona et al., 2015). At the end of the activity, each child will receive a sticker for their participation. The program has been gradually constructed using scientific evidence and is designed for one classroom period (15 minutes of instructions and closing, and 30 of direct play). All the activities are games with the following structure: an introduction with instructions and protagonist selection (an avatar who talks directly to the child and whose hair color, skin color, and clothes can be modified), followed by a practice exercise to ensure that the children understand what participants have to do (the exercise is repeated until the child performs it correctly), and, finally, the activity itself (4 different activities with 5 tries each). The first 10 sessions jointly stimulate working memory and emotion knowledge (4 activities focused on each skill per session), while the 10 remaining sessions stimulate inhibitory control and the selection of prosocial behaviors. The activities were constructed in previous projects by experts belonging to the research team. For example, in the working memory activities, the children receive phonological and visuo-spatial information and must recall this information in the same order that it was provided; in the inhibitory control activities, children must suppress automatic stimuli and processes; in the emotion recognition activities, kids must identify basic emotions; and in the selection of prosocial behaviors, and must choose an option to deal with a social problem. The intervention program covers some key ideas that any educational intervention aimed at preschoolers must consider a) Development and difficulty level: the activities will be structured from least to most difficult (a gradual approach to guarantee that all children will have a development-appropriate goal throughout the program; b) Variety of activities: each session features different activities; c) Short duration: the activities are short and dynamic; d) Achievable success: the program is constructed so that all children can succeed in their first attempts; e) Accessible and comprehensible instructions, with pertinent feedback (simple explanations with age-appropriate vocabulary and concepts); f) combination of play, practice, and learning (must have a ludic component, enabling children to practice until participants understand what must do before consolidating learning).

In this group, the educators will take part in 2 training sessions lasting 2 hours each in order to become familiar with the cognitive (working memory and inhibitory control), emotional (emotion recognition), and social skills (selection of prosocial behaviors) stimulated by the game, the functioning of the game, and its implementation in the classroom. Also, a meeting with all the educators will be held every 15 days to solve any doubts and evaluate the progression of the programs.

-Comparison group (active): The children will not work with the program for stimulating cognitive and socioemotional skills; however, over 20 sessions lasting 30 minutes each, 2 times per week, participants will play a tablet-based painting game that involves no cognitive, emotional, or social competence stimulation. At the end of the activity, each child will receive a sticker for their participation. In this group, the educators will receive the same training in cognitive, emotional, and social competence skills delivered to the intervention group. Children will also be trained in the use of the painting game, with meetings being held every 15 days to solve any doubts that might emerge. The similar treatment received by both groups is aimed at preventing teacher-dependent effects of the program. This knowledge will remain in place in each school for future studies in this field. All groups will be guided by the preschool educator in charge of the class and all the students will work at the same time (each child will have an individual tablet with headphones). All the children who wish to play will be able to participate (to avoid discrimination), however, only those who have their parents' consent and have given their assent will be able to do so. A member of the research team will be present in each session to ensure that it progresses adequately.

Instruments:

Each participant will be individually evaluated 6 times, 1 time before the intervention and 5 times after the intervention, using tasks focused on working memory, inhibitory control, emotion recognition, selection of prosocial behaviors, and pre-calculation and early literacy learning skills in 2 sessions lasting approximately 40 minutes each (with breaks throughout). The tasks will be administered at each school, in a quiet and controlled area. For their part, in the first months of each year, the parents will complete a questionnaire on the child's mental health (three times in total). The instruments used in the measurements were selected because: 1) tests have already been validated in Chile for small children (4 and 5 years of age) or are in the process of being validated by the team behind the present project, and 2) are in Spanish, are easy to use for small children, and are employed in research around the world.

Primary outcomes:

1- Tests of academic skills: 1.1- Initial literacy learning: Two tests will be used: Texas Lee, designed by the Texas Education Agency (2009) in collaboration with the University of Houston to evaluate reading in Spanish-speaking children. To evaluate vocabulary, the Spanish adaptation of the Kaufman Assessment Battery for Children (K-ABC) (Kaufman & Kaufman, 1997) will be used. Both were validated in Chile by Medina et al. (2011).

1.2- Pre-calculation skills: Woodcock-Muñoz (Battery III, Muñoz-Sandoval et al., 2005).

Control variable:

2. Mental health problems: Goodman's "Strengths and Difficulties Questionnaire" (SDQ) (1997) will be utilized. The version for children and young people in Chile was validated by some members of the present project (Gaete et al., 2018).

Potential mediators:

3. Tests of cognitive skills: 3.1. Working memory: For the visuo-spatial area, the "Corsi Cube test" (Corsi, 1972) will be administered. For the phonological area, the auditive memory subtest of Woodcock-Muñoz (Battery III, Muñoz-Sandoval et al., 2005) (internal consistency .80, Cizek, 2003) will be employed.

3.2 Inhibitory control: the "Hearts & Flowers" task (Diamond et al., 2007) will be used.

4. Tests of socio-emotional skills: 4.1. Emotion recognition: the "Assessment of Children's Emotional Skills" (ACES) by Shultz et al. (2004) will be administered. The test comprises 3 subscales: facial expressions, social situations, and social behavior. In the present project, the subscale of facial expressions (a =.68, Shultz et al., 2004) will be administered.

4.2 Selection of prosocial behaviors: the "Challenging Situations Task" (CST) by Denham et al. (1994) will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Establishments with an index of school vulnerability (ISV) ≥70%. (Based on information provided by participating families).
* Establishment that offers preschool and elementary education.
* Establishment located in the region of Maule, Chile.
* Co-educational School.
* Classes with a minimum of 15 students each.

Exclusion Criteria:

* School is implementing a similar program.
* Special education school.
* Children with a reported cognitive disability

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 754 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Texas Lee Test (Initial literacy learning) | 1 month
  An instrument designed to evaluate Initial literacy learning in Spanish-speaking children, validated for Chile and which considers the following dimensions: Book and Print Awareness (10 items), Phonological Awareness (12 items), Graphophonemic and phonological Knowledge (44 items), and Listening Comprehension (6 items). This test was designed for K1 to 3rd grade students.
Kaufman Assessment Battery for Children (K-ABC) (Vocabulary) | 1 month
  A measure of cognitive skill and academic knowledge used to evaluate the knowledge acquired and the level of school learning attained. This test was designed to evaluate children from 2 and a half to 12 and a half years old, in 4 dimensions: mental, sequential and simultaneous processing, and knowledge. The last one is the one will be used to measure vocabulary by 17 items.
subtest Battery III of Woodcock-Muñoz (Pre-calculation) | 1 month
  Pre-calculation skills using Battery III of Woodcock-Muñoz, which includes the following subtests: number identification (17 items), quantification (7 items), verbal counting (1 item), and applied problems (34 items). This test can be used to measure people from 5 to 95 years old.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) (Mental health problems) | 1 month
  A questionnaire comprising a set of emotional and behavioral problems experienced by children aged 4-16 years. It has 4 scales of psychological difficulties (with 5 items each): emotional symptoms, behavioral problems, hyperactivity/attention problems, problems among peers, and prosocial behavior.
Corsi Cube test (Visuo-spatial working memory) | 1 month
  This test requires repeating a sequence of up to nine identical blocks spatially separated on a screen which must be memorized for a short time to be repeated in the same order they were presented before or in the inverse order. The sequence is initially simple, but becomes more complex until the subject's performance starts decreasing. The test finishes if 2 consecutive errors are made in the same stage.
subtest of Battery III of Woodcock-Muñoz (Phonological working memory) | 1 month
  This test has 21 audio messages which contain numbers and words increasing the quantity and difficulty from lower to higher. Students are asked to remember and repeat these messages, if they fail 3 consecutive times the test ends.
Hearts & Flowers (Inhibitory control) | 1 month
  The task is a hybrid, combining elements from Simon and spatial tasks by Stroop, and contains congruent and incongruent trials which are organized in 3 parts and has a mean of 7 minutes of total duration.
Assessment of Children's Emotional Skills (ACES) (Emotion recognition) | 1 month
  The test comprises 3 subscales: facial expressions, social situations, and social behavior. In the present project, we will administer the subscale of facial expressions with 34 items in total. Students must recognize different emotions in photographs of school-age children.
Challenging Situations Task (CST) (Ability to select prosocial behaviors) | 1 month
  The instrument evaluates children's problem-solving skills. The participants will be shown 6 problems among peers and then the question "how would you feel?" being able to answer "happy", "sad", "mad", or "just fine" and mention what they would do. Their responses will be classified in four choices: prosocial, aggressive, crying, or avoidant.

IPD SHARING:
Plan to Share IPD: No
No share of individual participant data is planned because of restrictions provided by the Ethical Committee.

REFERENCES:
- [Background] Corsi, P. M. (1972). Human memory and the medial temporal region of the brain. Dissertation Abstracts International, 34 (2), 819B.
- [Background] Denham, S. A., Bouril, B., & Belouad, F. (1994). Preschoolers' affect and cognition about challenging peer situations. Child Study Journal, 24, 1-21.
- [Background] Diamond A, Barnett WS, Thomas J, Munro S. Preschool program improves cognitive control. Science. 2007 Nov 30;318(5855):1387-8. doi: 10.1126/science.1151148. PMID 18048670
- [Background] Gaete J, Montero-Marin J, Valenzuela D, Rojas-Barahona CA, Olivares E, Araya R. Mental health among children and adolescents: Construct validity, reliability, and parent-adolescent agreement on the 'Strengths and Difficulties Questionnaire' in Chile. PLoS One. 2018 Feb 5;13(2):e0191809. doi: 10.1371/journal.pone.0191809. eCollection 2018. PMID 29401472
- [Background] Kaufman, A. y Kaufman, N. (1997). Batería de Evaluación de Kaufman para niños k - abc. Madrid, España: TEA Ediciones
- [Background] Medina, L., Villalón, M., Meneses, A., Valdivia, A., Ruiz, M., San Martín, E., Förster, C., Martinic, S., & Cisterna, T. (2011). Alfabetización en establecimientos chilenos subvencionados. Informe final. Santiago de Chile: Ministerio de Educación.
- [Background] Muñoz-Sandoval, A. F., Woodcock, R. W., McGrew, K. S., & Mather, N. (2005). Batería III Woodcock-Muñoz. Itasca, IL: Riverside Publishing.
- [Background] Schultz D, Izard CE, Bear G. Children's emotion processing: relations to emotionality and aggression. Dev Psychopathol. 2004 Spring;16(2):371-87. doi: 10.1017/s0954579404044566. PMID 15487601
- [Background] Texas Education Agency (2009). Texas Reading First Initiative, 2008-2009 Commissioner's List of Reading Instruments. Recuperada el 18 de enero de 2010, http://ritter.tea.state.tx.us/curriculum/readingfirst/
- [Result] Blewitt C, Fuller-Tyszkiewicz M, Nolan A, Bergmeier H, Vicary D, Huang T, McCabe P, McKay T, Skouteris H. Social and Emotional Learning Associated With Universal Curriculum-Based Interventions in Early Childhood Education and Care Centers: A Systematic Review and Meta-analysis. JAMA Netw Open. 2018 Dec 7;1(8):e185727. doi: 10.1001/jamanetworkopen.2018.5727. PMID 30646283
- [Result] Herodotou, C. (2017). Young children and tablets: A systematic review of effects on learning and development. Journal of Computer Assisted Learning, 34, 1-9.
- [Result] Klingberg T, Fernell E, Olesen PJ, Johnson M, Gustafsson P, Dahlstrom K, Gillberg CG, Forssberg H, Westerberg H. Computerized training of working memory in children with ADHD--a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2005 Feb;44(2):177-86. doi: 10.1097/00004583-200502000-00010. PMID 15689731
- [Result] Rojas-Barahona, C. A., Förster Marín, C. E., Aboitiz, F., & Gaete, J. (2021). Are there differences in the development of the executive functions of children with a typical and atypical development stimulated by a game on a tablet? In C. Pracana & M. Wang (Eds.), Psychological Applications and Trends (pp. 349-353). Lisboa, Portugal: inScience Press
- [Result] Rojas-Barahona, C. A., Förster Marín, C. E., Moreno-Ríos, S., & McClelland, M. M. (2015). Improvement of Working Memory in Preschoolers and Its Impact on Early Literacy Skills: A Study in Deprived Communities of Rural and Urban Areas. Early Education & Development, 26(5-6), 871-892. doi: http://dx.doi.org/10.1080/10409289.2015.1036346.
- [Result] St. Clair-Thompson, H., Stevens, R., Hunt, A., & Bolder, E. (2010). Improving children's working memory and classroom performance. Educational Psychology, 30(2), 203-219
- [Derived] Rojas-Barahona CA, Gaete J, Veliz M, Castillo RD, Ramirez S, Araya R. The effectiveness of a tablet-based video game that stimulates cognitive, emotional, and social skills in developing academic skills among preschoolers: study protocol for a randomized controlled trial. Trials. 2022 Nov 9;23(1):936. doi: 10.1186/s13063-022-06875-9. PMID 36352445